CLINICAL TRIAL: NCT00165672
Title: A Clinical Pharmacology Study of E3810 With Pre- and Post-Treatment pH Monitoring in Patients With Non-Erosive Gastroesophageal Reflux Disease
Brief Title: A Study of E3810 With Pre- and Post-Treatment pH Monitoring in Patients With Non-Erosive Gastroesophageal Reflux Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Eisai Limited (Industry)
Responsible Party: Nobuyuki Sugisaki, Eisai Co., Ltd.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E3810-J081-462
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Results first posted 2011-10-05 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2010-08

CONDITIONS: Non-erosive Gastroesophageal Reflux Disease
Keywords: 24-hour esophageal pH monitoring; non-erosive gastroesophageal reflux disease; NERD; proton pump inhibitor; rabeprazole
MeSH Terms: interventions — Rabeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: RABEPRAZOLE SODIUM
- 2 (Experimental)
  Interventions: Drug: RABEPRAZOLE SODIUM

INTERVENTIONS:
Drug: RABEPRAZOLE SODIUM — rabeprazole sodium 5 mg: once daily orally for 4 weeks
  Arms: 1
Drug: RABEPRAZOLE SODIUM — rabeprazole sodium 10 mg: once daily orally for 4 weeks
  Arms: 2

SUMMARY:
To investigate esophageal reflux condition in patients with non-erosive gastroesophageal reflux disease by assessing with a 24-hour esophageal pH monitoring or effects of a 4-week treatment with 5 mg/day or 10 mg/day of E3810 (Pariet (Rabeprazole Sodium)).

ELIGIBILITY:
Inclusion Criteria:

The patients to be included will be outpatients who meet all of the following criteria. No specific gender is asked.

<For the observation period>

1. Patients who have "heartburn" 2 days a week or more during consecutive 3 weeks* prior to pre-observation screening. *If a day of screening and a day of starting observation (date of registration) are different, heartburn must continuously be present during the in-between period.
2. Patients who meet both 1) and 2) below;

1) The symptom is a burning sensation arising from the stomach or the lower chest.

2) The symptom tends to appear frequently or is aggravated after eating, when bending a body forward, and/or when pressing on the abdomen.

3. Patients categorized in "grade M" (discoloring type: minimal change) according to the Los Angeles System (2nd Modification) for Classification of Reflux Esophagitis.

4. Patients who are 20 years old or older at the time of obtaining consent.

5. Patients who are informed of the objective and details of this study and give written consent for study entry.

<For the treatment period>

1. Patients who have "heartburn" 2 days a week or more during 7 days until the treatment period (during the observation period).
2. Patients with "heartburn diary" that is completely filled out during 7 days until the treatment period (during the observation period). If the observation period is 8 days or longer, those with a heartburn diary of which entries are fulfilled 80% or more during the observation period.
3. Patients with 80% or better drug compliance for antacids during the observation period.
4. Patients whose percentage of time showing pH<4.0 (% time pH<4.0) is not 0%* during the 24-hour esophageal pH monitoring at the end of observation period (at the beginning of treatment period). *If parameters calculated from analytical program show 0.0% after round-off, this patient cannot be entered into the treatment period.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study.

1. Patients who cannot keep adequate entries of a heartburn diary by themselves.
2. Patients who strongly complain "feeling of heavy stomach" and/or "abdominal bloating."
3. Patients who have a complication or history of psychiatric or psychosomatic disease (e.g., manic-depressive psychosis, obsessive-compulsive neurosis, or others) or those who are on an antidepressant or anti-anxiety agent (accepted if only for a hypnotic treatment).
4. Patients who have undergone Helicobacter pylori eradication therapy, and less than 6 months* have elapsed from the end of H. pylori eradication therapy to the beginning of the observation period. *: The same day 6 months earlier, and the day at the end of 6 months earlier if it is at the end of month.
5. Patients with open gastric or duodenal ulcer.
6. Patients with acute gastritis.
7. Patients with a history of any surgical intervention that affect peptic secretion (e.g., upper gastrointestinal tract resection and/or vagotomy).
8. Patients with Barrett's esophagus, esophageal stenosis, or pyloric stenosis.
9. Patients with scleroderma.
10. Patients with a history or complication of angina pectoris.
11. Patients who work at night (working for a night-shift).
12. Patients who received proton pump inhibitors (PPIs) within 3 weeks prior to pre-observation screening.
13. Patients who need non steroidal anti-inflammatory drugs (NSAIDs) (except topical preparations), steroids (except topical preparations), and/or aspirin treatment every day.
14. Patients receiving dialysis therapy.
15. Patients with a serious complication such as cardiovascular disease (myocardial infarction, etc.), hematological disorder (e.g, aplastic anemia), renal disease (e.g., acute or chronic renal failure), hepatic disease (e.g., cirrhosis), or malignant tumor.
16. Patients with known hypersensitivity to antacids or PPIs.
17. Patients who are pregnant or those with childbearing potential, or those who wish to become pregnant or are lactating during the study period.
18. Patients receiving another investigational drug or those who received another investigational drug within 6 months prior to pre-observation screening* *: Registration is allowed on the same day of 6 months earlier, and the day at the end of 6 months earlier if it is at the end of month.
19. Patients who are judged to be ineligible for the study entry by the investigator or subinvestigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-05; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nobuyuki Sugisaki, Study Director — Eisai Co., Ltd - Development Clinical Research Department. Clinical Research Center
Locations (11):
- Japan (11):
  - Nagoya, Aichi-ken
  - Fukuoka, Fukuoka
  - Yukuhashi, Fukuoka
  - Hiroshima, Hiroshima
  - Osaka, Osaka
  - Saga, Saga-ken
  - Ōtsu, Shiga
  - Izumo, Shimane
  - Bunkyo-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Ube, Yamaguchi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 13 centers in Japan during the period of May-2005 to Oct-2005.
Pre-assignment Details: Antacid was administered 1-2 weeks for observational period (non-blind). Patients showing the resistance to antacid and patients for whom percent time with pH <4.0 >0% during the 24 hour esophageal pH monitoring at the end of the observation period.
Groups:
- E3810 Pariet (Rabeprazole Sodium) 5 mg: E3810 5 mg: once daily orally for 4 weeks
- E3810 Pariet (Rabeprazole Sodium) 10 mg: E3810 10 mg: once daily orally for 4 weeks
Period: Overall Study
Arm/Group | E3810 Pariet (Rabeprazole Sodium) 5 mg | E3810 Pariet (Rabeprazole Sodium) 10 mg
Started | 13 | 13
Completed | 13 | 12
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | E3810 Pariet (Rabeprazole Sodium) 5 mg | E3810 Pariet (Rabeprazole Sodium) 10 mg | Total
Number analyzed (Participants) | 9 | 9 | 18
Age Continuous [Mean (Standard Deviation); unit: years] — This number is the population for data analysis of clinical pharmacology.
  years | 40.6 (20.0) | 42.7 (15.8) | 41.6 (17.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 6 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Asian | 9 | 9 | 18
Region of Enrollment [Number; unit: participants]
  Japan | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: The Percent Time With pH <4.0 During 24 Hour Esophageal pH Monitoring at the End of the Observation Period (Predose Monitoring) and at the End of the Treatment Period (Postdose Monitoring).
Description: Mean and standard deviation of percent time pH<4.0 on 24 hour esophageal pH monitoring.
Time Frame: Baseline and 4 weeks
Population: The major endpoint of this study was analysed in the population for clinical pharmacology data (observation period and treatment period)
Measure: Mean (Standard Deviation); unit: Percent Time
Arm/Group | E3810 Pariet (Rabeprazole Sodium) 5 mg | E3810 Pariet (Rabeprazole Sodium) 10 mg
Number analyzed (Participants) | 9 | 9
Percent Time
  Baseline | 6.72 (5.30) | 7.03 (4.76)
  4 weeks | 1.38 (0.79) | 0.87 (1.22)

ADVERSE EVENTS:
Arm/Group | E3810 Pariet (Rabeprazole Sodium) 5 mg | E3810 Pariet (Rabeprazole Sodium) 10 mg
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 6/13 | 10/13
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E3810 Pariet (Rabeprazole Sodium) 5 mg (N=13) | E3810 Pariet (Rabeprazole Sodium) 10 mg (N=13)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Early satiety (General disorders) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No